CLINICAL TRIAL: NCT01857115
Title: A MULTICENTER, OPEN LABEL STUDY OF WEEKLY CARFILZOMIB, CYCLOPHOSPHAMIDE AND DEXAMETHASONE (wCCyd) IN NEWLY DIAGNOSED MULTIPLE MYELOMA (MM) PATIENTS
Brief Title: Study of Weekly Carfilzomib, Cyclophosphamide and Dexamethasone In Newly Diagnosed Multiple Myeloma Patients (wCCyd)
Acronym: wCCyd
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-CAR-561
Record Dates: First submitted 2013-04-17; First posted 2013-05-20 (Estimated); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Diagnosis; Weekly; CCyd
MeSH Terms: conditions — Multiple Myeloma; Disease | interventions — carfilzomib; Cyclophosphamide; Dexamethasone; Calcium Dobesilate

ARMS (1):
- CCyd (Experimental): Treatment schedule for 9 cycles of induction:
  1. Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15.
  2. Dexamethasone given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9,15-16, 22-23.
  3. Carfilzomib given 20 mg/m2 IV once daily on Day 1 of Cycle 1 only followed by 36/45/56/70 mg/m2 on days 8, 15 of Cycle 1, then for all subsequent doses 70 mg/m2 IV once daily on days 1, 8, 15, followed by 14-day rest period (day 16 through 28).
  Treatment schedule for maintenance until progression or intolerance:
  Carfilzomib at the MTD defined by phase I study IV once daily on days 1, 8, 15.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib
  Other Names: Krypolis
Drug: Cyclophosphamide
  Other Names: Endoxan
Drug: Dexamethasone
  Other Names: Decadron

SUMMARY:
This protocol is a phase I/II multicenter study designed to assess the safety and the efficacy of the proposed combinations as up-front treatment in elderly Multiple Myeloma (MM) patients.

DETAILED DESCRIPTION:
TREATMENT PERIOD Patients will start the induction treatment with wCCyd, as soon as the screening visits of the pre-treatment period have been terminated.

Each cycle will be repeated every 28 days for a total of 9 courses.

Treatment schedule for 9 cycles of induction:

Phase I:

In the phase I part of the study, the following dose levels of carfilzomib will be studied with constant doses of dexamethasone and cyclophosphamide to define the maximum tolerated dose (MTD):

Level -1

1. Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15.
2. Dexamethasone given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9,15-16, 22-23.
3. Carfilzomib given 20 mg/m2 IV once daily on Day 1 of Cycle 1 only followed by 36 mg/m2 on days 8, 15 of Cycle 1, then for all subsequent doses 36 mg/m2 IV once daily on days 1, 8, 15, followed by 14-day rest period (day 16 through 28).

Level 0 (starting dose)

1. Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15.
2. Dexamethasone given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9,15-16, 22-23.
3. Carfilzomib given 20 mg/m2 IV once daily on Day 1 of Cycle 1 only followed by 45 mg/m2 on days 8, 15 of Cycle 1, then for all subsequent doses 45 mg/m2 IV once daily on days 1, 8, 15, followed by 14-day rest period (day 16 through 28).

Level +1

1. Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15.
2. Dexamethasone given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9,15-16, 22-23.
3. Carfilzomib given 20 mg/m2 IV once daily on Day 1 of Cycle 1 only followed by 56 mg/m2 on days 8, 15 of Cycle 1, then for all subsequent doses 56 mg/m2 IV once daily on days 1, 8, 15, followed by 14-day rest period (day 16 through 28).

Level +2

1. Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15.
2. Dexamethasone given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9,15-16, 22-23.
3. Carfilzomib given 20 mg/m2 IV once daily on Day 1 of Cycle 1 only followed by 70 mg/m2 on days 8, 15 of Cycle 1, then for all subsequent doses 70 mg/m2 IV once daily on days 1, 8, 15, followed by 14-day rest period (day 16 through 28).

Patients will be observed during the first cycle of therapy for the assessment of side effects and observation of DLTs. Dose escalation will proceed as follows:

* 3 patients will be entered at dose level 0.
* If 0/3 patients experience DLT, dose escalation will continue.
* If 1/3 patients experience DLT, 3 additional patients will be added to this cohort (max 6).
* If no further patients experience DLT (1/6) dose escalation will continue.
* If 2/6 patients experience DLT, the MTD will have been exceeded and the MTD will be the previous dose at which < 2/6 experienced DLT.
* If 2/3 patients experience a DLT at any given dose, the MTD will have been exceeded and the MTD will be the preceding dose at which < 2/6 (or 1/3) patients experienced a DLT.

Phase II:

The dose used to treat patients in the phase II will be the MTD defined in the phase I of the study.

MAINTENANCE PERIOD At the end of the induction phase, patients will start the maintenance phase with Carfilzomib at the MTD defined by the phase I study IV once daily on days 1, 8, 15 until progression or intolerance.

Treatment schedule for maintenance until progression or intolerance:

Carfilzomib at the MTD defined by phase I study IV once daily on days 1, 8, 15.

ELIGIBILITY:
Inclusion Criteria:

Disease-related

1. Patient is a newly diagnosed MM patient.
2. Patient is age ≥ 65 year of age or who are ineligible for autologous stem cell transplantation.
3. Patient has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, ≥ 0.5 g/dL of M-protein) and, where applicable, urine light-chain excretion of > 200 mg/24 hours. For patients with oligo- or non-secretory MM, it is required that they have measurable plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan) or an abnormal free light chain ratio (n.v.: 0.26-1.65). We anticipate that less than 10% of patients admitted to this study will be oligo- or non-secretory MM with free light chains only in order to maximize interpretation of benefit results.

   Demographic:
4. Age ≥ 18 years.
5. Life expectancy ≥ 3 months.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Appendix F).

   Laboratory:
7. Adequate hepatic function, with serum ALT ≤ 3.5 times the upper limit of normal and serum direct bilirubin ≤ 2 mg/dL (34 µmol/L) within 14 days prior to randomization.
8. Absolute neutrophil count (ANC) ≥ 1.0 × 109/L within 14 days prior to randomization.
9. Corrected serum calcium ≤ 14 mg/dL (3.5 mmol/L).
10. Alanine transaminase (ALT): ≤ 3 x the ULN.
11. Hemoglobin ≥ 8 g/dL (80 g/L) within 14 days prior to randomization (subjects may be receiving red blood cell [RBC] transfusions in accordance with institutional guidelines).
12. Platelet count ≥ 50 × 109/L (≥ 30 × 109/L if myeloma involvement in the bone marrow is > 50%) within 14 days prior to randomization.
13. Creatinine clearance (CrCl) ≥ 15 mL/minute within 7 days prior to randomization, either measured or calculated using a standard formula (eg, Cockcroft and Gault).

    Ethical/Other:
14. Written informed consent in accordance with federal, local, and institutional guidelines.
15. Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing and to practice contraception.
16. Male subjects must agree to practice contraception.

Exclusion Criteria:

Disease-related:

1. Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid; ≤ to the equivalent of dexamethasone 40 mg/day for 4 days)
2. Patient with relapsed or refractory multiple myeloma.
3. Patients with non-secretory MM unless serum free light chains are present and the ratio is abnormal.

   Concurrent Conditions:
4. Pregnant or lactating females (Appendix I).
5. Major surgery within 21 days prior to randomization.
6. Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to randomization.
7. Known human immunodeficiency virus infection.
8. Active hepatitis B or C infection.
9. Unstable angina or myocardial infarction within 4 months prior to randomization, NYHA Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker.
10. Uncontrolled hypertension, uncontrolled congestive heart failure (CHF) or uncontrolled diabetes within 14 days prior to randomization.
11. Non-hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas.
12. Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to randomization.
13. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
14. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment.
15. Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to randomization.
16. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Identification of Dose-limiting toxicity (DLT) | 1 year
  Non-hematologic:
  * Grade2 neuropathy with pain
  * any Grade 3 toxicity (excluding nausea, vomiting, diarrhea)
  * Grade3 nausea, vomiting, or diarrhea despite maximal antiemetic/antidiarrheal therapy
  * Grade4 fatigue lasting for ≥7days
    * Any non-hematologic toxicity requiring a dose reduction within Cycle1
    * Inability to receive Day 1 dose of Cycle2 due to drug related toxicity persisting from Cycle1 or drug related toxicity newly encountered on Day1 of Cycle2.
  Hematologic:
  * Grade 4 neutropenia (ANC<0.5x109/L) lasting for ≥7days
  * Febrile neutropenia (ANC<1.0x109/L with a fever ≥38.3ºC)
  * Grade 4 thrombocytopenia (platelets<25.0x109/L) lasting ≥7 days despite dose delay
  * Grade 3-4 thrombocytopenia associated with bleeding
  * Any hematologic toxicity requiring a dose reduction within Cycle1
  * Inability to receive Day1 dose of Cycle2 due to drug related toxicity persisting from Cycle1 or drug related toxicity newly encountered on Day1 of Cycle2.
Partial Response (PR) | 1 year
  The primary efficacy endpoints will be assessed by considering partial response (PR) following the proposed regimen, at the end of third cycle.

SECONDARY OUTCOMES:
Response rate (RR) | 3 years
  Determine the response rate
Progression free-survival (PFS) | 3 years
  Determine progression free-survival
Time to progression (TTP) | 3 years
  Determine the time to progression
Duration of response (DOR) | 3 years
  Determine the duration of response
Overall survival (OS) | 3 years
  Determine the overall survival
Time to next therapy (TTNT) | 3 years
  Determine the time to next therapy
Responses | 3 years
  Determine whether responses obtained with wCCyd treatment are associated with a prolongation of PFS, in comparison with non-responding patients
Response and survival | 3 years
  Determine whether tumor response and survival might significantly change in particular subgroups of patients defined on prognostic factors (β2-microglobulin, C-reactive protein (CRP), FISH, gene expression profile)
Maintenance | 3 years
  * Determine the benefit on PFS and OS of maintenance with Carfilzomib
  * Determine the benefit on tumor load of maintenance with Carfilzomib

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione EMN Italy Onlus, Torino, Italy

REFERENCES:
- [Derived] Mina R, Bonello F, Petrucci MT, Liberati AM, Conticello C, Ballanti S, Musto P, Olivieri A, Benevolo G, Capra A, Gilestro M, Galieni P, Cavo M, Siniscalchi A, Palumbo A, Montefusco V, Gaidano G, Omede P, Boccadoro M, Bringhen S. Carfilzomib, cyclophosphamide and dexamethasone for newly diagnosed, high-risk myeloma patients not eligible for transplant: a pooled analysis of two studies. Haematologica. 2021 Apr 1;106(4):1079-1085. doi: 10.3324/haematol.2019.243428. PMID 32107329
- [Derived] Montefusco V, Gay F, Spada S, De Paoli L, Di Raimondo F, Ribolla R, Musolino C, Patriarca F, Musto P, Galieni P, Ballanti S, Nozzoli C, Cascavilla N, Ben-Yehuda D, Nagler A, Hajek R, Offidani M, Liberati AM, Sonneveld P, Cavo M, Corradini P, Boccadoro M. Outcome of paraosseous extra-medullary disease in newly diagnosed multiple myeloma patients treated with new drugs. Haematologica. 2020 Jan;105(1):193-200. doi: 10.3324/haematol.2019.219139. Epub 2019 Jun 20. PMID 31221778